CLINICAL TRIAL: NCT04133376
Title: The Effects of Electronic Hookah on Endothelial Cell Function: The Role of Nicotine
Brief Title: Electronic Hookah and Endothelial Cell Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Principal Investigator, Mary Rezk-Hanna, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: T30IP1013
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Smoking; Endothelial Dysfunction
MeSH Terms: conditions — Smoking | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-hookah vaping with nicotine (Experimental): Participants were invited to vape a 30-minute electronic hookah with nicotine vaping session, followed by a 30-minute electronic hookah without nicotine vaping session.
  To mitigate the impact of carryover effects, the two sessions were separated by a minimum of 7-days.
  Interventions: Other: Electronic hookah vaping with nicotine; Other: Electronic hookah vaping without nicotine
- e-hookah vaping without nicotine (Experimental): Participants were invited to vape a 30-minute electronic hookah without nicotine vaping session, followed by a 30-minute electronic hookah with nicotine vaping session.
  To mitigate the impact of carryover effects, the two sessions were separated by a minimum of 7-days.
  Interventions: Other: Electronic hookah vaping with nicotine; Other: Electronic hookah vaping without nicotine

INTERVENTIONS:
Other: Electronic hookah vaping with nicotine — Participants will be invited to vape a 30-minute session of e-hookah containing nicotine
Other: Electronic hookah vaping without nicotine — Participants will be invited to vape a 30-minute session of e-hookah without containing nicotine

SUMMARY:
Electronic nicotine delivery systems (ENDS) are a rapidly growing global epidemic among adolescents and young adults. Unlike other ENDS such as e-cigarettes, e-hookahs are used through traditional water-pipes, allowing the vapor-containing nicotine, propylene glycol, glycerin, and flavorings-to pass through a water-filled basin, potentially altering the vapor, before it is inhaled through the user's mouth. Contributing to e-hookahs popularity is the belief that the flavored smoke is detoxified as it passes through the water-filled basin, rendering e-hookah a safer tobacco alternative. However, an e-hookahs deliver flavored nicotine by creating a vapor of fine particles and volatile organic compounds that could induce vascular toxicity. While e-hookah vaping acutely reduces endothelial function, the specific role of nicotine and the mechanisms by which it may impairs endothelial function remain understudied. The objective of this project is to investigate the specific role of nicotine in mediating the acute effects of e-hookah vaping on endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* 21-39 years old hookah smokers: smoked hookah >12x in last 12 months
* 21-39 years old e-cigarette users: vaped >12x in last 12 months
* no history of illicit drugs
* no evidence of cardiopulmonary disease by history/ physical
* no diabetes: fasting blood glucose <100 mg/dl
* BP<140/90mmHg
* resting HR<100 bpm
* BMI<30kg•m2
* no prescription medication

Exclusion Criteria:

* exhaled CO>10 ppm (smoking non-abstinence)
* positive pregnancy test
* psychiatric illness

Ages: 21 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Flow-Mediated Dilation (FMD) | Changes pre- and post- the 30-minute smoking or vaping exposure sessions
  Using ultrasound, FMD of the brachial artery induced by reactive hyperemia, was used to measure endothelium-dependent vasodilator function. Outcome variable reflecting FMD (brachial artery diameter) was recorded for 45 seconds and resumed 30 seconds before cuff deflation and continuously for 2 minutes after deflation to obtain true peak vasodilatory response.
Acetylcholine-stimulated nitric oxide production | Changes pre- and post- the 30-minute smoking or vaping exposure sessions
  Human umbilical vein endothelial cells were cultured with subjects' serum sampled before and after the vaping sessions and acetylcholine-stimulated nitric oxide production was assessed
Basal reactive oxygen species bioactivity | Changes pre- and post- the 30-minute smoking or vaping exposure sessions
  Human umbilical vein endothelial cells were cultured with participants' serum sampled before and after the vaping sessions and basal reactive oxygen species bioactivity was assessed
Fibrinogen levels | Changes pre- and post- the 30-minute smoking or vaping exposure sessions
  Plasma fibrinogen
Heme oxygenase-1 assay | Changes pre- and post- the 30-minute smoking or vaping exposure sessions
  Heme oxygenase-1 concentration assay
paraoxonase-1 activity | Changes pre- and post- the 30-minute smoking or vaping exposure sessions
  paraoxonase-1 activity
HDL protection assay | Changes pre- and post- the 30-minute smoking or vaping exposure sessions
  HDL protection assay, reflecting the ability of HDL to inhibit oxidation to LDL
Nicotine levels | Changes pre- and post- the 30-minute smoking or vaping exposure sessions
  Plasma nicotine
Carbon monoxide levels | Changes pre- and post- the 30-minute smoking or vaping exposure sessions
  Exhaled carbon monoxide levels

CONTACTS AND LOCATIONS:
Overall Officials: Mary Rezk-Hanna, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided